CLINICAL TRIAL: NCT01249183
Title: An Open-label, Randomised, Multicentre Study to Evaluate the Immunogenicity and Safety of a Booster Dose of Diphtheria, Tetanus, Acellular Pertussis and Inactivated Poliomyelitis Adsorbed Vaccine (REPEVAX) Administered Concomitantly Versus Non-concomitantly With an Influenza Vaccine (VAXIGRIP) to Subjects of 60 Years of Age and Older
Brief Title: Safety and Immunogenicity Study of Concomitant Versus Non Concomitant Administration of a Diphtheria, Tetanus, Pertussis and Poliomyelitis Vaccine (REPEVAX) and Influenza Vaccine (VAXIGRIP) in Subjects Aged From 60 Years Old
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RPV03C
Record Dates: First submitted 2010-11-17; First posted 2010-11-29 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Diphtheria; Tetanus; Pertussis; Poliomyelitis
Keywords: Diphtheria; Tetanus; Pertussis (acellular, component); Diphteria; Biological / vaccine
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1- VAXIGRIP and REPEVAX concomitantly (Experimental)
  Interventions: Biological: Concomitant administration
- 2-REPEVAX 28 days after VAXIGRIP (Active Comparator)
  Interventions: Biological: Separate administration

INTERVENTIONS:
Biological: Concomitant administration — 1 dose (0.5 mL) of VAXIGRIP and 1 dose (0.5 mL) of REPEVAX in 2 separate injections sites (1 on each arm)
  Arms: 1- VAXIGRIP and REPEVAX concomitantly
Biological: Separate administration — 1 dose (0.5 mL) of VAXIGRIP at Day 0 and 1 dose (0.5 mL) of REPEVAX 28 days later
  Arms: 2-REPEVAX 28 days after VAXIGRIP

SUMMARY:
Primary objectives:

To demonstrate that REPEVAX and VAXIGRIP administered concomitantly in subjects 60 years of age and older are at least as immunogenic as REPEVAX or VAXIGRIP administered separately.

Secondary objectives:

•Secondary immunogenicity objectives: To describe the immune responses 28 days after concomitant or separate administration of REPEVAX and VAXIGRIP in subjects 60 years of age and older To describe the immune response of VAXIGRIP according to European Medicines Agency criteria in subjects 60 years of age and older (Note for Guidance, 1997: 28)

•Secondary safety objective: To describe the safety profile after vaccination in each group

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥60 years
* At least one documented booster dose with a tetanus- and diphtheria-containing vaccine between 5 and 15 years
* No influenza vaccine administered during the last 6 months

Exclusion Criteria:

* Receipt of a booster dose with a tetanus or diphtheria- or poliomyelitis- containing vaccine within the last 5 years
* Receipt of pertussis-containing vaccine or pertussis disease within the last 10 years
* Receipt of medication / vaccine that may interfere with study assessments
* Febrile illness or moderate or severe acute illness/infection
* History of hypersensitivity or anaphylactic or other allergic reactions to any of the vaccine components, or history of a life-threatening reaction to the study vaccines or a vaccine containing any of the same substances
* History of Guillain Barré syndrome or brachial neuritis following a previous vaccination
* History of encephalopathy of unknown origin within 7 days after immunization with a pertussis-containing vaccine or unstable neurological disorders
* Known or suspected immune dysfunction
* Thrombocytopenia, bleeding disorder or anticoagulants contraindicating intramuscular vaccination
* Chronic disease that is unstable or any intercurrent illness that might interfere with the ability to participate fully in the study; or interfere with evaluation of the vaccine

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 954 (Actual)
Dates: Start 2010-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Diphtheria seroprotection rate | 28 to 35 days after vaccine administration
Tetanus seroprotection rate | 28 to 35 days after vaccine administration
Polio seroprotection rate | 28 to 35 days after vaccine administration
Pertussis antibody titre | 28 to 35 days after vaccine administration
Flu geometric mean of titres ratio | 28 to 35 days after vaccine administration

SECONDARY OUTCOMES:
Solicited injection-site reactions, solicited systemic adverse reactions | From Day 0 to Day 7 following REPEVAX vaccination
Unsolicited injection-site adverse reactions and systemic adverse events | From Day 0 to Day 28 following REPEVAX and/or VAXIGRIP vaccination
Number and proportion of Serious adverse events | From the first visit to the last visit of the subject

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (20):
- France (12):
  - Sanofi Pasteur MSD Investigational Site, Angers
  - Sanofi Pasteur MSD Investigational Site, Châtellerault
  - Sanofi Pasteur MSD Investigational Site, Clermont-Ferrand
  - Sanofi Pasteur MSD Investigational Site, Gières
  - Sanofi Pasteur MSD Investigational Site, Grenoble
  - Sanofi Pasteur MSD Investigational Site, Hérouville-Saint-Clair
  - Sanofi Pasteur MSD Investigational Site, La Rochelle
  - Sanofi Pasteur MSD Investigational Site, Lyon
  - Sanofi Pasteur MSD Investigational Site, Poitiers
  - Sanofi Pasteur MSD Investigational Site, Strasbourg
  - Sanofi Pasteur MSD Investigational Site, Tiercé
  - Sanofi Pasteur MSD Investigational Site, Tours
- Germany (8):
  - Sanofi Pasteur MSD Investigational Site, Berlin
  - Sanofi Pasteur MSD Investigational Site, Dresden
  - Sanofi Pasteur MSD Investigational Site, Essen
  - Sanofi Pasteur MSD Investigational Site, Hamburg
  - Sanofi Pasteur MSD Investigational Site, Heilbronn
  - Sanofi Pasteur MSD Investigational Site, Künzing
  - Sanofi Pasteur MSD Investigational Site, Potsdam
  - Sanofi Pasteur MSD Investigational Site, Reichenbach